CLINICAL TRIAL: NCT01667588
Title: Sleep Disorders in Pediatric Dialysis
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Reshma Amin, Staff Respirologist, The Hospital for Sick Children
Other Study IDs: 1000031590
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Kidney Disease (CKD)
Keywords: Chronic Kidney Disease (CKD); Pediatrics; Sleep Disorders
MeSH Terms: conditions — Renal Insufficiency, Chronic; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre-Dialysis
- Dialysis

SUMMARY:
Sleep disorders (SD) are common in adults with Chronic Kidney Disease (CKD) on dialysis with a reported prevalence of 60-80%. To date three studies have reported on SDs in children with CKD but these have all been based on questionnaire data alone. The findings were not confirmed with polysomnograms (PSG), the gold standard to diagnose SD, or actigraphy, a validated tool to assess the sleep/ wake cycle over a prolonged period in the home. This is highly relevant given the poor sensitivity and specificity of even validated questionnaires alone. The effect of untreated pediatric SD is pervasive. This study will provide the first objective assessment of SDs using PSGs in children with severe CKD, both on and off dialysis. Therefore, we will recognize and when possible treat SD in this severe CKD cohort potentially contributing to their immediate management (eg improved control of hypertension, improved school performance), while improving their Quality of Life (QOL) and helping ensure they achieve their full potential.

ELIGIBILITY:
Inclusion Criteria:

* 0 to 18 years
* Caregivers must be able to read English
* Patients with either Stage 4 Chronic Kidney Disease (CKD) with an estimated GFR of 15-30 ml/min/1.73m2 based on IDMS Schwartz GFR OR patients with CKD receiving outpatient hemodialysis (HD) or peritoneal dialysis (PD) for a minimum of 1 month
* Informed consent

Exclusion Criteria:

* Caregivers cannot read English
* Informed consent not given

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The two study cohorts will be age and sex matched and constructed as follows:
  1. Pre-dialysis: Stage 4 CKD with an estimated GFR of 15-30 ml/min/1.73m2 based on IDMS Schwartz GFR
  2. Dialysis: CKD receiving outpatient hemodialysis (HD) or peritoneal dialysis (PD) for a minimum of 1 month. The PSG will be completed after the longest inter-dialytic interval for HD patients. Patients on PD will undergo PSG while on their usual cycler nocturnal dialysis regimen.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2012-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of Sleep Disorders | Baseline
  Report the prevalence of sleep disorders in a cohort of severe Chronic Kidney Disorder children both on and off dialysis based on PSG, actigraphy, and questionnaire.

SECONDARY OUTCOMES:
Quality of Life | Baseline
  The Pediatric Quality of Life Inventory (Peds QL) generic core (version 4.0) scale is a 23-item multidimensional instrument for measuring pediatric HRQL.

CONTACTS AND LOCATIONS:
Overall Officials: Reshma Amin, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada